CLINICAL TRIAL: NCT01548131
Title: A Randomized Longitudinal Trial About Treatment for Severe Fear of Childbirth
Acronym: LINNEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Hanna Rouhe, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 228/2006
Record Dates: First submitted 2012-02-18; First posted 2012-03-08 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Fear of Childbirth
Keywords: fear of childbirth; delivery mode; delivery satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychoeducative group therapy (Experimental): Psychoeducative group therapy
  Interventions: Behavioral: Psychoeducative group therapy
- Control (No Intervention): Women screened for fear of childbirth were taken cared by primary health care nurses and if needed referred to specialized care in hospital
  Interventions: Behavioral: Psychoeducative group therapy

INTERVENTIONS:
Behavioral: Psychoeducative group therapy — 6 sessions during pregnancy and 1 after childbirth

SUMMARY:
Site of research: Helsinki University Central Hospital (HUCH), Department of Obstetrics and Gynaecology and University of Helsinki Department of Psychology, in collaboration with Karolinska University Hospital in Stockholm, Sweden

In Finland and in Sweden, fear of childbirth is one of the most common reasons for consultation of obstetrician, and for an elective caesarean section. Approximately 5 to 6% of pregnant women suffer from severe fear of childbirth, which disturbs family-life and working and prevents the preparation to normal childbirth and parenthood. It represents as nightmares, panic attacks, anxiety, and as numerous physical complaints. After giving birth it can be difficult for these women to form an early mother-infant-relationship. Their risk for puerperal depression is also increased.

Finland and Sweden have both a long tradition in research of this field. In Finland, the investigators research group started the first out-patient clinic for fearful pregnant women in HUCH in1996. Different strategies how to treat fear of childbirth have been applied to clinical practise. Studies on the treatment for fear of childbirth are, however, scanty. Some descriptive studies have showed that far more than one half of patients can, after the treatment, prepare to a normal vaginal delivery and caesarean without a medical indication can be avoided. The aim of the treatment should be both to avoid unnecessary caesareans, increase the number of uneventful vaginal deliveries and to help the pregnant couple to prepare to parenthood, as well as to prevent puerperal depression.

In this study, psychotherapeutic group psychoeducation is studied as promising treatment for severe fear of childbirth. To screen fear of childbirth, all women coming to ultrasound screening at the 18 to 20 gestational week in HUCH are asked to fill in a specific questionnaire. Those nulliparous women whose score for fear exceeds 95th percentile are randomized to intervention and to control group.

The intervention group is invited to start a psychotherapeutic group therapy based on cognitive and psychodynamic therapy combined with training in relaxation. Each group consists of six nulliparous women and meets six times during pregnancy 120 minutes at a time. Between the sessions the patients fill in a homework questionnaire. One session focuses on the partner's role and the partners are present then. Three months after delivery, the groups meet once more.

The women in the control group stay in the care of community midwives and general physicians. If needed, they are referred to out-patient clinic in the maternity hospital where their fear is treated according the clinical practice of that hospital, mainly support from obstetrician or midwife.

The women and their partners in both groups are asked, approximately one month after the screening and one month before the due date of delivery, to fill in the questionnaires examining depression, self-esteem, general anxiety, social support, marital satisfaction, personal projects and concerns, and efficacy concerning childbirth and maternity. After childbirth, data about the childbirth will be collected. Three months and two years after childbirth mothers and fathers in both groups receive again a psychosocial questionnaires.

The aim of the study is to help the authorities to organize the treatment for fear of childbirth in their districts by examining the benefits of the treatment also in long-run. The investigators hope the results would lead to production of Current Care guidelines for fear of childbirth.

ELIGIBILITY:
Inclusion Criteria:

* severe fear of childbirth

Exclusion Criteria:

* twin pregnancies

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2007-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
number of spontaneous vaginal deliveries | after delivery within a month
  delivery information is collected from patient records after delivery

SECONDARY OUTCOMES:
specific questionnaires about mental wellbeing | two years after delivery
  two time-points: three months after delivery and two years after delivery
specific questionnaire about delivery satisfaction | three months after delivery
specific questionnaire about early mother-infant-relationship | three months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Terhi Saisto, MD, PhD, Study Director — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, HUS, Finland

REFERENCES:
- [Derived] O'Connell MA, Khashan AS, Leahy-Warren P, Stewart F, O'Neill SM. Interventions for fear of childbirth including tocophobia. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013321. doi: 10.1002/14651858.CD013321.pub2. PMID 34231203